CLINICAL TRIAL: NCT03653793
Title: LivRelief Varicose Veins Cream in the Treatment of Chronic Venous Insufficiency of the Lower Limbs: A 6-week Single Arm Pilot Study
Brief Title: LivRelief Varicose Veins Cream in the Treatment of Varicose Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delivra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020990
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Intervention Model Description: This was a single arm pilot study to determine the feasibility of conducting an appropriately sized RCT within the same population using the same clinical outcome measures.
  Eligible adult patients of the clinic with varicose veins were asked to use the cream as directed on the packaging for 6-weeks and the post-treatment measures were compared to baseline data. This study also provided SDs of the sample for comparison to the study population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LivRelief Varicose Veins Cream (Experimental): Intervention:
  All subjects were provided with an adequate supply of the Natural Health Product LivRelief Varicose Veins cream for 6 weeks of at home use.
  Interventions: Other: Natural Health Product: LivRelief Varicose Veins Cream

INTERVENTIONS:
Other: Natural Health Product: LivRelief Varicose Veins Cream — This product is intended to improve circulation and blood flow to minimize the appearance of varicose veins.
  Other Names: Natural Product Number (NPN) 80029349

SUMMARY:
Phase IV interventional design where all participants used the test product as per package instructions for 6-weeks. Baseline observations were compared to those collected after 6-weeks of treatment.

DETAILED DESCRIPTION:
The use of the marketed natural product, LivRelief Varicose Veins Cream, was observed in 32 patients with lower limb varicose veins. Participants were recruited from the patient population at The Mayer Institute in Hamilton Ontario, Canada. Patients that agreed to participate in the study and met the eligibility criteria were provided with a 6-week supply of the cream to use at home as directed on the product packaging. The following study measures were performed at the clinic prior to the first use of the cream, then again at the clinic after 6 weeks of use: CEAP (Clinical, Etiological, Anatomical, Pathophysiological) classification and VCSS (Venous Clinical Severity score). These are assessments performed by the doctor or nurse to determine the severity of their varicose veins and CVI (chronic venous insufficiency), measurements taken of the circumference of their legs to measure swelling of the legs, photographs of the varicose veins, a quality of life enjoyment and satisfaction questionnaire (QLES-Q-SF) completed by the subjects to describe their satisfaction with various aspects of their life over the last week and documentation of any reactions to the treatment. The cream was applied to their varicose veins twice a day for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years of age.
* Presence of lower limb varicose veins.

Exclusion Criteria:

* Allergy to witch-hazel or any allergies in the cream.
* Intent to undergo surgical treatment varicose veins within the next six weeks.
* Pregnant or breastfeeding or planning to be pregnant.
* Any Dementia or Major Cognitive dysfunction that would preclude the individual's ability to provide informed consent or complete the Case Report Form.
* Any unstable medical condition (including but not limited to cardiovascular, cardiac/hypertension disease, moderate to severe kidney disease, and moderate to severe liver disease)
* Any medical condition that would preclude the participant's or a caregiver's ability to administer the product on a daily basis for the time period required to complete the study.
* An active ulcer at the site of product application (as evaluated during CEAP screening).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | study duration:~4 weeks
  Recruitment of at least 70% of all eligible participants
Data Collection | study duration: ~6 to 12 weeks
  Collection of at least 70% of scheduled data

CONTACTS AND LOCATIONS:
Overall Officials: Perry V Mayer, MD, Principal Investigator — The Mayer Institute
Locations (1):
- The Mayer Institute, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dwyer HC, Baranowski DC, Mayer PV, Gabriele S. LivRelief varicose veins cream in the treatment of chronic venous insufficiency of the lower limbs: A 6-week single arm pilot study. PLoS One. 2018 Dec 31;13(12):e0208954. doi: 10.1371/journal.pone.0208954. eCollection 2018. PMID 30596677